CLINICAL TRIAL: NCT04545060
Title: A Phase II/III Randomized, Multi-center, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of Monoclonal Antibody VIR-7831 for the Early Treatment of Coronavirus Disease 2019 (COVID-19) in Non-hospitalized Patients
Brief Title: VIR-7831 for the Early Treatment of COVID-19 in Outpatients
Acronym: COMET-ICE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIR-7831-5001; GSK Study 214367 (Other: GlaxoSmithKline)
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Covid19
Keywords: SARS-CoV-2; coronavirus; coronavirus disease 2019; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — sotrovimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIR-7831 (Sotrovimab) (Experimental): Participants received 500 mg sotrovimab administered intravenously (IV)
  Interventions: Biological: VIR-7831 (sotrovimab)
- Placebo (Placebo Comparator): Participants received placebo administered intravenously (IV)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: VIR-7831 (sotrovimab) — VIR-7831 (sotrovimab) given by intravenous infusion (single dose)
  Arms: VIR-7831 (Sotrovimab)
Drug: Placebo — Sterile normal saline (0.9% NaCl) given by intravenous infusion (single dose)
  Arms: Placebo

SUMMARY:
This is a phase 2/3 study in which subjects with coronavirus disease 2019 (COVID-19) will receive VIR-7831 or placebo and will be assessed for safety, tolerability, efficacy, and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be aged 18 years or older AND at high risk of progression of COVID-19 or ≥ 55 years old
* Participants must have a positive SARS-CoV-2 test result and oxygen saturation ≥94% on room air and have COVID-19 symptoms and be less than or equal to 5 days from onset of symptoms

Exclusion Criteria:

* Currently hospitalized or judged by the investigator as likely to require hospitalization in the next 24 hours
* Symptoms consistent with severe COVID-19
* Participants who, in the judgement of the investigator are likely to die in the next 7 days
* Severely immunocompromised participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (78):
- United States (52):
  - Investigative Site, Anniston, Alabama
  - Investigative Site, Cullman, Alabama
  - Investigative Site, Mesa, Arizona
  - Investigative Site, Tucson, Arizona
  - Investigative Site, Los Angeles, California
  - Investigative Site, Northridge, California
  - Investigative Site, Oxnard, California
  - Investigative Site, Rolling Hills Estates, California
  - Investigative Site, Sacramento, California
  - Investigative Site, Doral, Florida
  - Investigative Site, Gainesville, Florida
  - Investigative Site, Hialeah, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Miramar, Florida
  - Investigative Site, North Miami, Florida
  - Investigative Site, Palmetto Bay, Florida
  - Investigative Site, Pembroke Pines, Florida
  - Investigative Site, Pompano Beach, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Decatur, Georgia
  - Investigative Site, Stockbridge, Georgia
  - Investigative Site, Idaho Falls, Idaho
  - Investigative Site, Mishawaka, Indiana
  - Investigative Site, Lake Charles, Louisiana
  - Investigative Site, Marrero, Louisiana
  - Investigative Site, Baltimore, Maryland
  - Investigative Site, Caro, Michigan
  - Investigative Site, Hazelwood, Missouri
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, Santa Fe, New Mexico
  - Investigative Site, The Bronx, New York
  - Investigative Site, Asheboro, North Carolina
  - Investigative Site, Charlotte, North Carolina
  - Investigative Site, Columbus, Ohio
  - Investigative Site, Smithfield, Pennsylvania
  - Investigative Site, Chattanooga, Tennessee
  - Investigative Site, Austin, Texas
  - Investigative Site, Baytown, Texas
  - Investigative Site, Beaumont, Texas
  - Investigative Site, Dallas, Texas
  - Investigative Site, Denton, Texas
  - Investigative Site, El Paso, Texas
  - Investigative Site, Forney, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, Humble, Texas
  - Investigative Site, Laredo, Texas
  - Investigative Site, McAllen, Texas
  - Investigative Site, Mesquite, Texas
  - Investigative Site, Sugar Land, Texas
  - Investigative Site, Kirkland, Washington
  - Investigative Site, Seattle, Washington
- Investigative Site, Vienna, Austria
- Brazil (9):
  - Investigative Site, Belo Horizonte, Minas Gerais
  - Investigative Site, Maringá, Paraná
  - Investigative Site, Natal, Rio Grande do Norte
  - Investigative Site, Passo Fundo, Rio Grande do Sul
  - Investigative Site, Porto Alegre, Rio Grande do Sul
  - Investigative Site, Chapecó, Santa Catarina
  - Investigative Site, Campinas, São Paulo
  - Investigative Site, Santo André, São Paulo
  - Investigative Site, Vila Assuncao, São Paulo
- Canada (3):
  - Investigative Site, Sarnia, Ontario
  - Investigative Site, Toronto, Ontario
  - Investigative Site, Québec, Quebec
- Peru (6):
  - Investigative Site, El Agustino, Lima region
  - Investigative Site, Huaral, Lima region
  - Investigative Site, San Isidro, Lima region
  - Investigative Site, Bellavista, Provincia Constitucional del Callao
  - Investigative Site, Bella Vista
  - Investigative Site, Lima
- Spain (6):
  - Investigative Site, Centelles, Barcelona
  - Investigative Site, Terrassa, Barcelona
  - Investigative Site, Albacete
  - Investigative Site, Girona
  - Investigative Site, Granada
  - Investigative Site, Vigo
- Investigative Site, Belfast, United Kingdom

REFERENCES:
- [Result] Maher MC, Soriaga LB, Gupta A, Chen YP, di Iulio J, Ledoux S, Smithey MJ, Cathcart AL, McKusick K, Sun D, Aldinger M, Alexander E, Purcell L, Ding X, Peppercorn A, Austin D, Mogalian E, Yeh WW, Shapiro AE, Corti D, Virgin HW, Pang PS, Telenti A. Antibody therapy reverses biological signatures of COVID-19 progression. Cell Rep Med. 2022 Aug 16;3(8):100721. doi: 10.1016/j.xcrm.2022.100721. PMID 35977462
- [Result] Gupta A, Gonzalez-Rojas Y, Juarez E, Crespo Casal M, Moya J, Rodrigues Falci D, Sarkis E, Solis J, Zheng H, Scott N, Cathcart AL, Parra S, Sager JE, Austin D, Peppercorn A, Alexander E, Yeh WW, Brinson C, Aldinger M, Shapiro AE; COMET-ICE Investigators. Effect of Sotrovimab on Hospitalization or Death Among High-risk Patients With Mild to Moderate COVID-19: A Randomized Clinical Trial. JAMA. 2022 Apr 5;327(13):1236-1246. doi: 10.1001/jama.2022.2832. PMID 35285853
- [Result] Gupta A, Gonzalez-Rojas Y, Juarez E, Crespo Casal M, Moya J, Falci DR, Sarkis E, Solis J, Zheng H, Scott N, Cathcart AL, Hebner CM, Sager J, Mogalian E, Tipple C, Peppercorn A, Alexander E, Pang PS, Free A, Brinson C, Aldinger M, Shapiro AE; COMET-ICE Investigators. Early Treatment for Covid-19 with SARS-CoV-2 Neutralizing Antibody Sotrovimab. N Engl J Med. 2021 Nov 18;385(21):1941-1950. doi: 10.1056/NEJMoa2107934. Epub 2021 Oct 27. PMID 34706189
- [Derived] Subramanian S, Schnell G, Iulio JD, Gupta AK, Shapiro AE, Sarkis EH, Lopuski A, Peppercorn A, Aldinger M, Hebner CM, Cathcart AL. Resistance analysis following sotrovimab treatment in participants with COVID-19 during the phase III COMET-ICE study. Future Virol. 2023 Nov:10.2217/fvl-2023-0146. doi: 10.2217/fvl-2023-0146. Epub 2023 Dec 7. PMID 38074312
- [Derived] Satram S, Ghafoori P, Reyes CM, Keeley TJH, Birch HJ, Brintziki D, Aldinger M, Alexander E, Lopuski A, Sarkis EH, Gupta A, Shapiro AE, Powers JH 3rd. Assessment of symptoms in COMET-ICE, a phase 2/3 study of sotrovimab for early treatment of non-hospitalized patients with COVID-19. J Patient Rep Outcomes. 2023 Sep 13;7(1):92. doi: 10.1186/s41687-023-00621-8. PMID 37702920
- [Derived] Keeley TJH, Satram S, Ghafoori P, Reyes C, Birch HJ, Raymond K, Gelhorn HL, Kosinski M, Saucier CD, Mitchell Foster A, Lopuski A, Powers JH 3rd. Content validity and psychometric properties of the inFLUenza Patient-Reported Outcome Plus (FLU-PRO Plus(c)) instrument in patients with COVID-19. Qual Life Res. 2023 Jun;32(6):1645-1657. doi: 10.1007/s11136-022-03336-3. Epub 2023 Jan 27. PMID 36703019
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised two parts: lead-in phase and expansion phase
Groups:
- Sotrovimab (500 mg IV): Participants received 500 mg sotrovimab administered intravenously (IV)
Period: Overall Study
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Started | 528 | 529
Completed | 498 | 488
Not Completed | 30 | 41
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 5
Not completed — Lost to Follow-up | 10 | 13
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 17 | 22

BASELINE CHARACTERISTICS:
Population: All participants who were randomly assigned to study intervention in the study ( irrespective of whether they have been dosed)
Groups:
- Total: Total of all reporting groups
Arm/Group | Sotrovimab (500 mg IV) | Placebo | Total
Number analyzed (Participants) | 528 | 529 | 1057
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 6
  Between 18 and 65 years | 421 | 417 | 838
  >=65 years | 105 | 108 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (15.07) | 52.6 (14.76) | 52.1 (14.92)
Age, Customized [Median (Full Range); unit: years] | 53 [18 to 96] | 53 [17 to 88] | 53 [17 to 96]
Age, Customized [Count of Participants; unit: Participants]
  Randomized Age Group Strata, Categorical: <=70 years | 472 | 473 | 945
  Randomized Age Group Strata, Categorical: >70 years | 56 | 56 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299 | 273 | 572
  Male | 229 | 256 | 485
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 345 | 346 | 691
  Not Hispanic or Latino | 183 | 183 | 366
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 24 | 21 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 42 | 82
  White | 458 | 463 | 921
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 479 | 474 | 953
  Canada | 24 | 28 | 52
  Spain | 14 | 15 | 29
  Brazil | 11 | 11 | 22
  Peru | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: kg] — Weight at Screening
  kg | 89.5 (21.5) | 90.05 (21.3) | 89.8 (21.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index at Screening
  kg/m^2 | 32.3 (6.7) | 32.2 (6.6) | 32.3 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Progression of COVID-19 Through Day 29
Description: COVID-19 progression defined as hospitalization >24 hours or death
Time Frame: Through Day 29
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 6 | 30
Statistical Analysis 1: Comparison: Sotrovimab (500 mg IV) vs Placebo; Test type: Superiority; p < 0.001, poisson regression model — two-sided, alpha=0.05; adjusted relative risk ratio = 0.21, 95% CI 2-sided [0.09 to 0.50]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Up to 24 weeks
Population: All participants who received at least one dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 523 | 526
Participants | 133 | 140

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Time Frame: Up to 24 weeks
Population: All participants who received at least one dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 523 | 526
Participants | 11 | 35

4. Secondary Outcome: Number of Participants With Infusion-related Reactions (IRR) Including Hypersensitivity Reactions
Time Frame: Up to 24 weeks
Population: All participants who received at least one dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 523 | 526
Participants | 7 | 6

5. Secondary Outcome: Number of Participants With Cardiac Events of Special Interest
Time Frame: Up to 24 weeks
Population: All participants who received at least one dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 523 | 526
Participants | 1 | 0

6. Secondary Outcome: Number of Participants With Serum Anti-drug Antibody (ADA) to Sotrovimab
Time Frame: Up to 24 weeks
Population: Number of subjects with any post-baseline ADA result
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 513 | 4
Participants | 65 | 0

7. Secondary Outcome: Titers of Serum Anti-drug Antibody (ADA) to Sotrovimab
Description: Titers defined as the reciprocal of the highest dilution of the sample (including minimum required dilution) that yields a positive result.
Time Frame: Up to 24 Weeks
Population: Safety (subjects with any post-baseline ADA)
Measure: Median (Full Range); unit: Titer
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 513 | 4
Titer
  Treatment-induced | 40 [10 to 1280] | 0 [0 to 0]
  Treatment-boosted | 80 [10 to 5120] | 0 [0 to 0]
  Treatment-unaffected | 10 [10 to 80] | 0 [0 to 0]

8. Secondary Outcome: Maximum Observed Concentration (Cmax) of VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: Participants in the Lead-in phase (n=10) who received 500 mg sotrovimab administered intravenously (IV). One subject was excluded from summary due to insufficient data (no data before study Day 5).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Sotrovimab 500 mg IV (Lead-In Phase): Participants in the Lead-in phase received 500 mg sotrovimab administered intravenously (IV)
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
μg/mL | 245.6 (39.44)

9. Secondary Outcome: Concentration at the Last Quantifiable Time Point (Clast) of VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: Participants in the Lead-in phase (n=10) who received 500 mg sotrovimab administered intravenously (IV). One subject was excluded from summary due to insufficient data (no data past study Day 2).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
μg/mL | 8.4 (44.41)

10. Secondary Outcome: Time to Reach the Maximum Concentration (Tmax) of VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 8
Measure: Median (Full Range); unit: day
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
day | 0.04 [0.04 to 0.05]

11. Secondary Outcome: Time of the Last Quantifiable Concentration (Tlast) of VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 9
Measure: Median (Full Range); unit: day
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
day | 161 [160 to 167]

12. Secondary Outcome: Area Under the Serum Concentration-time Curve Extrapolated From Zero to Infinity (AUCinf) of VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
day*μg/mL | 5536.9 (25.18)

13. Secondary Outcome: Area Under the Serum Concentration-time Curve From the Time of Dosing to the Time of the Last Measurable (Positive) Concentration (AUClast) of VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
day*μg/mL | 4777.7 (20.15)

14. Secondary Outcome: Percentage of AUCinf Obtained by Extrapolation (%AUCexp) for VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
percentage | 12.6 (41.26)

15. Secondary Outcome: Terminal Elimination Half-life (t1/2) of VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 9
Measure: Median (Full Range); unit: day
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
day | 56.5 [42.4 to 77.3]

16. Secondary Outcome: Apparent Volume of Distribution During the Elimination Phase (Vz) of VIR-7831 Following IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
Liter | 7.52 (13.77)

17. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of VIR-7831 Following IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
Liter | 6.93 (11.59)

18. Secondary Outcome: Clearance (CL) of VIR-7831 After IV Administration
Time Frame: Day 1: Pre-dose, and end of infusion; Days 2, 5, 8, 15, 29, 43, 57, 85, 141, 169
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | Sotrovimab 500 mg IV (Lead-In Phase)
Number analyzed (Participants) | 9
mL/day | 90.3 (25.18)

19. Secondary Outcome: Number of Participants Who Had Progression of COVID-19
Description: COVID-19 progression defined as a visit to a hospital emergency room for management of illness or hospitalization for acute management of illness or death
Time Frame: Through Day 29
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 13 | 39
Statistical Analysis 1: Comparison: Sotrovimab (500 mg IV) vs Placebo; Test type: Superiority; p < 0.001, poisson regression model — two-sided, alpha=0.05; relative risk ratio = 0.34, 95% CI 2-sided [0.19 to 0.63]

20. Secondary Outcome: Mean Change in FLU PRO Plus Total Score (AUC)
Description: Mean change in InFLUenza Patient-Reported Outcome (FLU-PRO Plus) questionnaire total score.
  The FLU-PRO is a 32-item daily diary assessing influenza symptoms and severity across 6 body systems (nose, throat, eyes, chest/respiratory, gastrointestinal, and body/systemic). The FLU-PRO Plus includes the 32-item FLU-PRO with 2 additional items for loss of smell and taste. The mean total score can range from 0 (symptom free) to 4 (very severe symptoms) and was calculated as the arithmetic mean of the 32 items within FLU-PRO. Missing total score at day 7 was imputed using a modified last observation carried forward approach.
Time Frame: Through Day 7
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention) with available FLU-PRO Plus total scores to calculate AUC through Day 7.
Measure: Least Squares Mean (95% Confidence Interval); unit: Total symptom score x days
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 412 | 399
Total symptom score x days | -3.05 [-3.27 to -2.83] | -1.98 [-2.20 to -1.76]
Statistical Analysis 1: Comparison: Sotrovimab (500 mg IV) vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — two-sided, alpha=0.05; Least squares mean difference = -1.07, 95% CI 2-sided [-1.38 to -0.76]

21. Secondary Outcome: Time to Symptom Alleviation Using FLU-PRO Plus
Description: Symptom alleviation is defined as absence of the majority of core symptoms of COVID-19 (except for cough or fatigue, where scoring no more than 'somewhat' in severity, and loss of smell or taste were allowed) as measured by FLU-PRO Plus, sustained for >=48 hours. Participants could only achieve sustained symptom alleviation following >=2 non-missing consecutively scored questionnaires that showed symptom alleviation. Participants who did not achieve sustained symptom alleviation were censored at Day 21, the day of death, or the day of withdrawal, whichever was earliest. Days where symptom alleviation could not be assessed to a missing/incomplete questionnaire were imputed as no symptom alleviation.
  The FLU-PRO is a 32-item daily diary assessing influenza symptoms and severity across 6 body systems (nose, throat, eyes, chest/respiratory, gastrointestinal, and body/systemic). The FLU-PRO Plus includes the 32-item FLU-PRO with 2 additional items for loss of smell and taste.
Time Frame: Through Day 21
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Number; unit: Days
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Days | NA — It was not possible to calculate the median time to sustained symptom alleviation due to the high proportion of missing data | NA — It was not possible to calculate the median time to sustained symptom alleviation due to the high proportion of missing data

22. Secondary Outcome: Change From Baseline in Viral Load in Nasal Secretions by qRT-PCR at Day 8
Time Frame: Baseline and Day 8
Population: Participants in the Virology analysis population (all participants who were randomly assigned to study intervention with a central lab confirmed quantifiable baseline nasopharyngeal swab) with analyzable data at Day 8
Measure: Least Squares Mean (Standard Error); unit: Log 10 copies/mL
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 294 | 305
Log 10 copies/mL | -2.589 (0.0606) | -2.357 (0.0598)
Statistical Analysis 1: Comparison: Sotrovimab (500 mg IV) vs Placebo; Test type: Superiority; p = 0.007, Mixed model repeated measures — two-sided, alpha=0.05; Least squares mean difference = -0.232, 95% CI 2-sided [-0.399 to -0.065]

23. Secondary Outcome: Number of Participants Who Progressed to Develop Severe and/or Critical Respiratory COVID-19 as Manifested by Requirement for and Method of Supplemental Oxygen Through Day 8
Time Frame: Through Day 8
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 6 | 20

24. Secondary Outcome: Number of Participants Who Progressed to Develop Severe and/or Critical Respiratory COVID-19 as Manifested by Requirement for and Method of Supplemental Oxygen Through Day 15
Description: Participants were defined as progression to severe respiratory COVID-19 if they required supplemental oxygen either by nasal cannula, face mask, high-flow oxygen devices, or non-invasive ventilation. Participants were defined as progression to critical respiratory COVID-19 if they required invasive mechanical ventilation or ECMO.
Time Frame: Through Day 15
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 6 | 28

25. Secondary Outcome: Number of Participants Who Progressed to Develop Severe and/or Critical Respiratory COVID-19 as Manifested by Requirement for and Method of Supplemental Oxygen Through Day 22
Description: as for outcome 24
Time Frame: Through Day 22
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 7 | 28

26. Secondary Outcome: Number of Participants Who Progressed to Develop Severe and/or Critical Respiratory COVID-19 as Manifested by Requirement for and Method of Supplemental Oxygen Through Day 29
Description: as for outcome 24
Time Frame: Through Day 29
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 7 | 28
Statistical Analysis 1: Comparison: Sotrovimab (500 mg IV) vs Placebo; Test type: Superiority; p = 0.002, poisson regression model — two-sided, alpha=0.05; relative risk ratio = 0.26, 95% CI 2-sided [0.12 to 0.59]

27. Secondary Outcome: 29-day All-cause Mortality
Description: Participants alive at the respective follow-up timepoint were censored at that timepoint; participants who withdrew prior to the respective timepoint were censored at the time of study withdrawal
Time Frame: Through Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 0 | 2

28. Secondary Outcome: 60-day All-cause Mortality
Description: as for outcome 27
Time Frame: Through Day 60
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 0 | 4

29. Secondary Outcome: 90-day All-cause Mortality
Description: as for outcome 27
Time Frame: Through Day 90
Population: Intent-to-Treat (All participants who were randomly assigned to study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab (500 mg IV) | Placebo
Number analyzed (Participants) | 528 | 529
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: Baseline Up to 24 Weeks
Description: All participants who received at least one dose of study intervention
Arm/Group | Sotrovimab (500 mg IV) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/523 | 5/526
Serious Adverse Events (participants affected / at risk) | 11/523 | 35/526
Other Adverse Events (participants affected / at risk) | 26/523 | 31/526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotrovimab (500 mg IV) (N=523) | Placebo (N=526)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 20 (20)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotrovimab (500 mg IV) (N=523) | Placebo (N=526)
Nausea (Gastrointestinal disorders) | 6 (6) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 4 (5)
Headache (Nervous system disorders) | 7 (8) | 11 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7)
Hypertension (Vascular disorders) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT04545060/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04545060/SAP_001.pdf